CLINICAL TRIAL: NCT06755268
Title: Effect of Music on Comfort, Anxiety and Hemodynamic Parameters During Coronary Angiography
Brief Title: Effect of Music on Coronary Angiography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Özlem Canbolat (Other)
Responsible Party: Sponsor-Investigator, Özlem Canbolat, Assistant Professor, Gazi University
Organization: Gazi University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-77082166-302.08.01-850481
Record Dates: First submitted 2024-09-24; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-07

CONDITIONS: Coronary Angiography; Hemodynamic Parameters; Comfort; Anxiety; Music Intervention
Keywords: Anxiety; Comfort; Coronary angiography; Hemodynamic parameters; Nursing
MeSH Terms: conditions — Anxiety Disorders | interventions — Wind; Walking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Application Group (Experimental): After explaining the purpose of the study and the way it was applied to patients in the music group, Introductory Information Form, State Anxiety Scale," "General Comfort Scale," and "Hemodynamic Parameters Record Form were applied. The intervention group listened to nature sounds (the sound of birds, water flowing in a river, wind or walking in the forest) based music during the angiography procedure.Music was played to the intervention group via a loudspeaker placed in the coronary angiography laboratory.The intervention group was reapplied the State Anxiety Scale, General Comfort Scale and Hemodynamic Parameters Record Form after the angiography procedure.
  Interventions: Other: listening to nature sounds (the sound of birds, water flowing in a river, wind or walking in the forest) based music
- Control Group (No Intervention): After explaining the purpose of the study and the way it was applied to patients in the control group, Introductory Information Form, State Anxiety Scale," "General Comfort Scale," and "Hemodynamic Parameters Record Form were applied. No application was be made to the control group. The control group was reapplied the State Anxiety Scale, General Comfort Scale and Hemodynamic Parameters Record Form after the angiography procedure.

INTERVENTIONS:
Other: listening to nature sounds (the sound of birds, water flowing in a river, wind or walking in the forest) based music — Listening to nature sounds (the sound of birds, water flowing in a river, wind or walking in the forest) based music during the angiography procedure.
  Arms: Application Group

SUMMARY:
This study was conducted in a randomized, controlled experimental design to examine the effect of music on comfort, anxiety and hemodynamic parameters during coronary angiography. The research was conducted with 78 patients (39 intervention and 39 control groups) who were processed in the Coronary Angiography Laboratory of Necmettin Erbakan Training and Research Hospital between February and June 2024. The intervention group listened to nature sounds based music during the angiography procedure, but no intervention was made to the control group. "Introductory Information Form," "State Anxiety Scale," "General Comfort Scale," and "Hemodynamic Parameters Record Form" were used to collect the data.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older
* Being at least literate
* Having no mental and cognitive competence
* Understanding and speaking Turkish
* Having a planned coronary angiography
* Performing for diagnostic purposes

Exclusion Criteria:

* Having visual and hearing impairment
* Having a psychiatric diagnosis
* Using psychiatric medication (tranquilizers, etc.)
* Using anxiety medication in the last 6 months
* Having had coronary angiography before
* The coronary angiography procedure is being performed for therapeutic purposes (stent, balloon, etc.)
* An unexpected complication during coronary angiography (arrhythmia, MI, bleeding, etc.)
* coronary angiographyprocedure started for diagnostic purposes and stent and/or balloon procedures were applied during the procedure
* Data collection forms were not filled out by the participant after coronary angiography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
General Comfort Scale | before the angiography procedure and after the angiography procedure (average of 15 minutes)
  Scores from the scale range from 48 to 192, and the higher the score, the higher the comfort level.

SECONDARY OUTCOMES:
State Anxiety Scale | before the angiography procedure and after the angiography procedure (average of 15 minutes)
  Scores from the scale range from 20 to 80, and the higher the score, the higher the anxiety level.

OTHER OUTCOMES:
Hemodynamic Parameters Record Form | before the angiography procedure and after the angiography procedure (average of 15 minutes)
  The form was used to record the Systolic Blood Pressure (mm/Hg), Diastolic Blood Pressure (mm/Hg), Respiratory Rate, Heart Rate (Pulse) (atm/min) and Saturation parameters measured before and after the angiography procedure of the intervention and control groups.
  Systolic blood pressure measurements were averaged. Diastolic blood pressure measurements were averaged. Saturation measurements were averaged. Respiratory rate measurements were averaged. Heart Rate (Pulse) measurements were averaged.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided